CLINICAL TRIAL: NCT05854758
Title: Effects of Core Strengthening on Mechanical Back Pain in Overweight Adults.
Brief Title: Effects of Core Strengthening on Mechanical Low Back Pain in Overweight Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01410 JUNAID UR RAHMAN
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Low Back Pain, Mechanical; Overweight
Keywords: low back pain; overweight; exercise; core strengthening; numerical pain rating scale
MeSH Terms: conditions — Low Back Pain; Overweight; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core strengthening with conventional treatment (Experimental): This group will perform planks, side planks and superman exercises along with knee to chest, pelvic rotation, back extension, and bridge exercises after baseline treatment of therapeutic hot pack and transcutaneous electrical nerve stimulation continuous mode for 10 minutes.
  Interventions: Other: Core strengthening with conventional treatment
- Conventional treatment (Active Comparator): This group will perform knee to chest, pelvic rotation, bridge and back extension exercises after baseline treatment of therapeutic hot pack and transcutaneous electrical nerve stimulation. continuous mode for 10 minutes. Each exercise will be repeated 10 times, with 10 second holds, followed by a five-minute rest interval
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Core strengthening with conventional treatment — A detailed musculoskeletal examination of lumbar spine will be performed before the start of treatment. Oswestry Low Back Pain Disability Questionnaire for pain will be noted. An expert physical therapist with more than 7 years clinical experience will assist the patients in performing core stabilization exercise with conventional physical therapy protocol and routine physical therapy exercise. The session with the physical therapist will usually last for up to 40 minutes.
  This group will perform planks, side planks and superman exercises along with knee to chest, pelvic rotation, back extension, and bridge exercises after baseline treatment of therapeutic hot pack and transcutaneous electrical nerve stimulation. continuous mode for 10 minutes.
  Arms: Core strengthening with conventional treatment
Other: Conventional treatment — A detailed musculoskeletal examination of lumbar spine will be performed before the start of treatment. Oswestry Low Back Pain Disability Questionnaire for pain will be noted. An expert physical therapist with more than 7 years clinical experience will assist the patients in performing core stabilization exercise with conventional physical therapy protocol and routine physical therapy exercise. The session with the physical therapist will usually last for up to 40 minutes.
  This group will perform knee to chest, pelvic rotation, bridge and back extension exercises after baseline treatment of therapeutic hot pack and transcutaneous electrical nerve stimulation. continuous mode for 10 minutes. Each exercise will be repeated 10 times, with 10 second holds, followed by a five-minute rest interval
  Arms: Conventional treatment

SUMMARY:
The goal of this clinical trial is to determine the effects of core strengthening on mechanical back pain in overweight adults.

The main question is aims to answer:

Is there an effect of core strengthening on mechanical back pain in overweight adults? The participants will be divided into two groups; group A and group B Group A will perform core strengthening after baseline treatment of therapeutic hot pack and Trans continuous mode for 10 minutes.

Group B will perform conventional exercises after baseline treatment of therapeutic hot pack and transcutaneous electrical nerve stimulation. continuous mode for 10 minutes. Each exercise will be repeated 10 times, with 10 second holds, followed by a five-minute rest interval.

DETAILED DESCRIPTION:
Low back pain (LBP) is defined as low back pain that keep on for more than 3 months, and it is the most commonly reported clinical symptom of orthopedic diseases. Low back pain has been the leading cause of disability globally for at least the past three decades and results in enormous direct healthcare and lost productivity costs. More than 50% of people in the United States are affected by LBP, and it is the primary cause of work nonappearance and everlasting disability. The core muscles, which are the primary muscle group for maintaining spinal strength, can be separated into two groups according to their functions and attributes.

The origin of LBP is complex, several of which are unidentified. Management of chronic low back pain (CLBP) is often multidisciplinary, involving a combination of treatments, including therapeutic exercises. Core stability exercises aim to improve pain and disability in CLBP increasing spinal stability, neuromuscular control, and preventing shear force that causes injury to the lumbar spine. One major cause involves the weakening of the shallow trunk and abdominal muscles. Another cause of CLBP is the deteriorating of or insufficient motor control of the deep trunk muscles, such as the lumbar multifidus and transversus abdominis. Lumbar multifidus (LM), the main trunk stabilization muscle, may have reduced efficiency 24 h after the onset of acute LBP.

During physical activities, the trunk muscle tissues ensure the mobility and stability of the lumbopelvic region; thus, changes in trunk muscle activity (particularly in the lumbar multifidus and transversus abdominis) are typically observed in patients with low back pain. Stabilization exercise programs have been widely applied for LBP treatment because they were effective in reducing LBP and disability. Core strength training is directed at working out the deep trunk muscles. However, autonomous training is challenging for LBP patients despite the existence of numerous core strength training strategies. Furthermore, no standardized system has been established for analyzing and comparing the results of core strength training and typical resistance training (6).

Core strengthening impression have gained increased popularity in low back rehabilitation. Traditional low back pain rehabilitation is based on a stationary spine stability model and is composed mostly of modalities, stretching and strengthening exercises (7). More recent theories, however, include newer concepts of dynamic spinal stability, coordination and neuromuscular control. Core strengthening exercises incorporate these new concepts. Although more research is required, the best available evidence suggests that a core strengthening program may be advantageous in reducing pain scores, functional disability and recurrences of acute low back pain episodes. Strong clinical and emerging epidemiological evidence shows that muscle-strengthening exercises is independently associated with multiple health outcomes, including a reduced risk of all-cause mortality, incidence of diabetes and enhanced metabolic , musculoskeletal and mental health.

Low back pain (LBP) is an economic burden to society, leading to functional disability resulting in loss of number of days at work. Literature review state that 75% or more patients with low back become temporarily disabled and around 5% people suffer from permanent disability .

Diagnosis of mechanical low back pain is commonly made by physical examination, physical tests, palpation, imaging such as x-rays, MRI, and CT scan. Medication, physical therapy, and surgery are most commonly used managements of mechanical low back pain. The physical therapy management varies according to the patient condition, and includes modalities, exercise therapy, manual therapy and patient's education with a comprehensive home plan of care.

The individual effectiveness of manual physical therapy and core stability exercises therapy are evident in the management of mechanical low back pain, but there is no single study available in the literature on the combined effects of physical therapy and core stability exercise therapy. The objective of the current study will be to determine the combined effect of physical therapy and core stability exercise therapy in the management of mechanical low back pain.

The conventional physical therapy is a commonly used management of mechanical low back pain to improve the mobility of the lumbar spine. The core stabilization exercises for strengthening of spinal muscles to improve their ability to maintain neutral spine using the abdominal, back, neck and shoulder girdle muscles as stabilizers rather than movers. Trunk stability exercises that focus on either deep or superficial muscles might produce different effects on lumbar segmental motion .

Obesity is a complex disease that accumulated excess body fat leads to negative effects on health.

Obesity persists to accelerate resulting in an unprecedented epidemic that shows no significant signs of slowing down any time soon. Raised body mass index (BMI) is a risk factor for illness such as diabetes, cardiovascular diseases, and musculoskeletal disorders, resulting in dramatic decrease of life quality and expectancy. The main cause of obesity is long-term energy imbalance between consumed calories and expended calories. Here, The purpose of our study is to find out the effect of core strengthening on LBP and total body fat.

ELIGIBILITY:
Inclusion Criteria:

* Males & Female
* Age: 25-45
* Chronic low back pain for more than 3 months .
* BMI of 25 or greater
* Body fat percentage > 25%
* Numerical Pain Rating Scale ratings less than 7

Exclusion Criteria:

Participant failing to fall in this category would be excluded of the study.

* Patients with non-mechanical low back pain
* Patients with acute low back pain.
* Post laminectomy/discectomy
* Spondylolisthesis
* Osteoporosis/Fractures
* Cauda equine syndrome
* Recent history of spinal trauma or surgery
* Lumbar myelopathy
* Patients with known metabolic diseases
* Patients with any neurological deficit

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-07-08 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | 6 weeks
  The 11-point Numerical Pain Rating Scale consists of numbers between 0 and 10 where 0 indicates "no pain" and 10 indicates "maximum pain." The respondent is instructed to identify one number between 0 and 10, which is best representative of their pain intensity
Oswestry Low Back Pain Disability Questionnaire | 6 weeks
  The Oswestry Disability Index (ODI) is one of the most commonly used outcome measures for individuals with low back pain. Psychometric properties of the ODI will determine the questionnaire's suitability as a useful clinical tool. The ODI is a valid, reliable, and responsive condition-specific assessment tool that is suited for use in clinical practice. It is easy to administer and score, objectifies clients' complaints, and monitors effects of therapy
Body Mass Index | 6 weeks
  Body Mass Index is a simple calculation using a person's height and weight. The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in meters squared. A BMI of 25.0 or more is overweight, while the healthy range is 18.5 to 24.9.
Total Body Fat | 6 weeks
  The Jackson-Pollack method for evaluating body fat percentage requires three skin fold measurements. For men, measurement sites are the chest, abdomen and thigh; for women, they consist of the thigh, triceps and suprailiac crest, or just above the top of the hip bone. Because measurements are taken in very specific spots, precise locations are typically measured and marked with a washable marker before the test is conducted. For consistency and accuracy, all skin fold measurements are taken at least twice on the right side of a standing, relaxed body and should never be taken after exercise, when a person's fluid levels can interfere with accuracy. Measurements are taken on the right side of body. Caliber needs to be perpendicular to the site analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Jawad Naweed, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- Elite Physical Therapy Centre, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No